CLINICAL TRIAL: NCT03629574
Title: Evaluation of a Protocol of Protective Mechanical Ventilation During Cardiopulmonary Bypass in Cardiosurgery for Congenital Heart Diseseas
Brief Title: Mechanical Ventilation During Cardiopulmonary Bypass
Acronym: VENICE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Cristiana Carollo, Medical Doctor, Azienda Ospedaliera di Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 34365
Record Dates: First submitted 2018-06-19; First posted 2018-08-14 (Actual); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Congenital Heart Disease; Mechanical Ventilation Complication; Cardiopulmonary Bypass
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilated Group (Experimental): This group will receive a protective mechanical ventilation during cardiopulmonary byass. No drugs will be administered.
  Interventions: Procedure: Ventilation during cardiopulmonary bypass
- Not-ventilated group (No Intervention): This group will not receive any kind of mechanical ventilation during cardiopulmonary byass. The ventilator will be switched off.

INTERVENTIONS:
Procedure: Ventilation during cardiopulmonary bypass — Mechanical ventilation during cardiopulmonary bypass
  Arms: Ventilated Group

SUMMARY:
The study is about a protocol of protective mechanical ventilation during cardiopulmonary bypass used during cardiosurgery for the correction of congenital heart diseases, to evaluate what's the best for the lungs

ELIGIBILITY:
Inclusion Criteria:

* congenital heart diseases
* younger than 5 years
* CPB longer than 30 minutes in hypotermia
* elective surgery
* stable clinical conditions

Exclusion Criteria:

* genetic anomalies
* mechanical ventilation before the surgery
* kidney injuries
* hepatic failure

Max Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2018-08-20 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the damage of the air-blood membrane in a ventilation protocol and a non ventilation protocol during cardiopulmonary bypass | Baseline, and 6, 12, 24 and 48 hours after the surgery
  It will be assed the plasma level of proteins which usually are absent in the plasma (surfactant protein A and B) that change as a damage of the air-blood membrane appears.

CONTACTS AND LOCATIONS:
Locations (1):
- AOPadova, Padua, Italy